CLINICAL TRIAL: NCT04677101
Title: Liquid Biopsy as a Non-invasive Tool for the Diagnosis of NASH and Liver Fibrosis
Brief Title: Liquid Biopsy for NASH and Liver Fibrosis
Acronym: LIBRA
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Professor, Catholic University of the Sacred Heart
Other Study IDs: 20201612
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; Liver Fibroses
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with NASH documented by liver biopsy: One hundred subjects with NASH documented by liver biopsy and no evidence of another form of liver disease with a BMI ≥30 and ≤55 kg/m2.
  Interventions: Diagnostic Test: Liver Biopsy
- Healhy Donor: Fifty subjects with normal liver who underwent laparoscopic elective cholecystectomy, but otherwise in healthy conditions, will be used as controls.
  Interventions: Diagnostic Test: Liver Biopsy

INTERVENTIONS:
Diagnostic Test: Liver Biopsy — Fine-needle liver biopsy

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) has evolved to represent the most common cause of chronic liver disease globally. Today, NAFLD is a leading indication for liver transplantation and a major etiology for hepatocellular carcinoma (HCC) in the United States. NAFLD is characterized by the excess accumulation of lipids within the liver and ranges from isolated steatosis to nonalcoholic steatohepatitis (NASH), which is characterized by the presence of hepatic necroinflammation, hepatocyte ballooning and fibrosis progression.

Currently, liver biopsy remains the gold standard for the diagnosis of various chronic liver diseases, and for determining the severity of liver injury, inflammation, and fibrosis stage. However, this procedure is invasive, prone to complications such as bleeding and is associated with sampling variability and limited representation of the whole liver. Other limitations include, the difficulty to monitor liver injury progression over time and underestimation of disease severity.

Despite intensive research, currently available non-invasive blood tests are not sufficiently sensitive or specific and are therefore of limited use. Blood biomarkers might provide significant advances in the diagnosis and monitoring of disease progression and regression in clinical settings.

Recently, liquid biopsy has emerged as a potential, less invasive, alternative to liver biopsy. In fact, it addresses several unmet clinical needs, including sensitivity, specificity, the determination of prognoses, and the prediction of therapeutic responses.

DETAILED DESCRIPTION:
This is a multicentric prospective observational study to validate blood non-invasive biomarkers for NASH and fibrosis stage.

150 subjects will be enrolled; 100 subjects with biopsy-proven NASH and 50 subjects with normal liver will be used as controls.

ELIGIBILITY:
Inclusion Criteria:

One hundred subjects with NASH documented by liver biopsy and no evidence of another form of liver disease with a BMI ≥30 and ≤55 kg/m2.

Fifty subjects with normal liver who underwent laparoscopic elective cholecystectomy, but otherwise in healthy conditions, will be used as controls.

Exclusion Criteria:

Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous 6 months; Liver cirrhosis; End stage renal failure; Participation in any other concurrent therapeutic clinical trial; Any other life-threatening, non-cardiac disease; Pregnancy; Inability to give informed consent; Substantial alcohol consumption (>20 g/day for women or >30 g/day for men); Wilson's disease; Lipodystrophy; Parenteral nutrition; Interfering medications (e.g., amiodarone, methotrexate, tamoxifen, corticosteroids).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: One hundred subjects with NASH documented by liver biopsy and no evidence of another form of liver disease with a BMI ≥30 and ≤55 kg/m2.
  Fifty subjects with normal liver who underwent laparoscopic elective cholecystectomy, but otherwise in healthy conditions, will be used as controls.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
The primary aim of our study is to validate blood non-invasivebiomarker sensitivity and accuracy in predicting NASH and fibrosis stage. | 2 months

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University of Rome Sapienza, Roma
  - Catholic University School of Medicine, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angelini G, Panunzi S, Castagneto-Gissey L, Pellicano F, De Gaetano A, Pompili M, Riccardi L, Garcovich M, Raffaelli M, Ciccoritti L, Verrastro O, Russo MF, Vecchio FM, Casella G, Casella-Mariolo J, Papa L, Marini PL, Rubino F, le Roux CW, Bornstein S, Mingrone G. Accurate liquid biopsy for the diagnosis of non-alcoholic steatohepatitis and liver fibrosis. Gut. 2023 Feb;72(2):392-403. doi: 10.1136/gutjnl-2022-327498. Epub 2022 Jul 12. PMID 35820779